CLINICAL TRIAL: NCT06459427
Title: Robot-Assisted Minimally Invasive Surgery for Brainstem Hemorrhage
Brief Title: A Multicenter, RAndomIzed, coNtrolled, umBrella Trial fOr Minimally Invasive Neurosurgery With AI-assisted Robotic guidanCe for Hemorrhagic Stroke
Acronym: RAINBOW-BSH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yanbing Yu (Other)
Responsible Party: Sponsor-Investigator, Yanbing Yu, Chief of Neurosurgery, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01084205031
Record Dates: First submitted 2024-06-06; First posted 2024-06-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Brain Stem Hemorrhage; Robotic Surgical Procedures
MeSH Terms: interventions — Nutrition Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted minimally invasive puncture and aspiration surgery (Experimental): The intervention group will receive robot-assisted stereotactic puncture for brainstem hemorrhage
  Interventions: Procedure: Robot-assisted minimally invasive puncture and aspiration surgery; Other: Standard medical management
- Standard medical management (Active Comparator): The control group will undergo conventional medical conservative management.
  Interventions: Other: Standard medical management

INTERVENTIONS:
Procedure: Robot-assisted minimally invasive puncture and aspiration surgery — Positioning and surgical operation will be performed according to the robot navigation system protocols. Preoperative imaging data will be used for precise surgical planning, including the construction of a three-dimensional (3D) preoperative visualization model. The 3D reconstruction and CT data will be imported into the AI robot-assisted stereotactic system, which, after mapping to the patient's skull, automatically designs the surgical target, calculates coordinate values, plans the puncture trajectory, and determines the cranial entry point. Different surgical approaches will be selected based on the location and shape of the hematoma, and individualized parameters, including puncture direction and trajectory length, will be generated for each patient. During the procedure, the robot will assist with stereotactic puncture, while the patient's heart rate and blood pressure are closely monitored.
  Other Names: Neurosurgical Robot
  Arms: Robot-assisted minimally invasive puncture and aspiration surgery
Other: Standard medical management — According to the "Chinese Neurosurgical Expert Consensus on the Diagnosis and Treatment of Primary Brainstem Hemorrhage", conventional medical treatment includes oxygen therapy, specialized nursing care, blood pressure control (maintaining BP at ≤140/90 mmHg), sedation, intracranial pressure reduction, arousal promotion, gastric protection, maintenance of internal homeostasis, infection prevention, neuro-nutrition, brain function support, nutritional support, and overall systemic management; For comatose patients, ensure a patent airway, provide nebulization and sputum clearance, prevent respiratory depression, and improve respiratory function. Closely monitor the patient's condition and provide active symptomatic treatment as needed. Regular cranial CT scans are performed to evaluate intracranial status, and in cases of ventricular hemorrhage or obstructive hydrocephalus, lateral ventricular puncture and drainage may be performed.
  Other Names: Medical therapy

SUMMARY:
The purpose of this clinical trial is to observe the improvements in clinical symptoms and imaging outcomes for brainstem hemorrhage using robot-assisted stereotactic puncture, evaluate the clinical efficacy and safety of this treatment, and explore the development of a high-precision, intelligent, and individualized microsurgical diagnosis and treatment process for brainstem hemorrhage. The main questions it aims to address are:

* Establish a multi-center clinical database for brainstem hemorrhage.
* Clinically observe and evaluate the intervention effects of robot-assisted stereotactic puncture on brainstem hemorrhage, compare it with the traditional conservative treatment control group, and investigate its efficacy and impact on patient survival, motor evoked potentials, and the degree of neurological deficits.
* Optimize the Artificial Intelligence (AI) algorithm-based robotic surgical assistance system, and explore the prediction of preoperative brainstem hematoma stability and hematoma path planning.

Participants in the experimental group will:

* Undergo robot-assisted stereotactic minimally invasive surgery for brainstem hematoma puncture
* Receive conservative non-surgical treatment.

If there is a control group: the researchers will compare the conservative non-surgical treatment group to evaluate the effectiveness of robot-assisted stereotactic minimally invasive surgery for brainstem hematoma puncture.

ELIGIBILITY:
Participants must meet all of the following inclusion criteria:

1. Age ≥18 years at randomization；
2. Diagnosed with brainstem hemorrhage via imaging (CT, CTA, etc.)；
3. Hematoma volume ≥3 mL；
4. Glasgow Coma Scale (GCS) score of 3-12；
5. Available for surgery within 48 hours after onset；
6. Modified Rankin Scale (mRS) score ≤ 1 prior to this hemorrhage；
7. Informed consent obtained in accordance with national laws, regulations, and applicable ethics committee requirements.

Patients will be excluded if they meet any of the following criteria:

1. Hematoma involving other regions such as the supratentorial compartment, basal ganglia, thalamus, midbrain, or ventricles.
2. Radiologically confirmed cerebral vascular abnormalities including ruptured aneurysms, arteriovenous malformations (AVMs), or Moyamoya disease; hemorrhagic transformation of ischemic infarcts; or recent (within 1 year) recurrence of intracerebral hemorrhage；
3. Any irreversible coagulation disorder or known coagulopathy; platelet count <100,000/µL; INR >1.4; or use of anticoagulant medication within 7 days before the current hemorrhage；
4. Current or probable pregnancy；
5. Patients with concurrent severe illness likely to influence outcome assessment；
6. Difficulty in follow-up or poor compliance due to any cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 60 days
  60 days survival rate after follow-up

SECONDARY OUTCOMES:
Ordinal shift in mRS scores at 60 days and 6 months | 60 days and 6 months
  The modified Rankin Scale (mRS) is a standardized tool used to assess the neurological recovery status of stroke patients. The scale is divided into seven levels, ranging from 0 to 6. Higher scores indicate more severe patient conditions.
Favorable functional outcome at 60 days and 6 months (mRS 0-1) | 60 days and 6 months
  The modified Rankin Scale (mRS) is a standardized tool used to assess the neurological recovery status of stroke patients. The scale is divided into seven levels, ranging from 0 to 6. Higher scores indicate more severe patient conditions.
Functional independence at 60 days and 6 months (mRS 0-2) | 60 days and 6 months
  The modified Rankin Scale (mRS) is a standardized tool used to assess the neurological recovery status of stroke patients. The scale is divided into seven levels, ranging from 0 to 6. Higher scores indicate more severe patient conditions.
Health-related quality of life (HRQoL) at 60 days and 6 months, assessed by the EQ-5D-5L questionnaire | 60 days and 6 months
  Health-related quality of life (HRQoL) at 60 days and 6 months, assessed by the EQ-5D-5L questionnaire
Utility-weighted mRS at 60 days and 6 months | 60 days and 6 months
  The modified Rankin Scale (mRS) is a standardized tool used to assess the neurological recovery status of stroke patients. The scale is divided into seven levels, ranging from 0 to 6. Higher scores indicate more severe patient conditions.
Cognitive function at 60 days and 6 months | 60 days and 6 months
  Cognitive function at 60 days and 6 months
Total length of hospital stay | 60 days
  Total length of hospital stay
Costs during hospitalization | 60 days
  Costs during hospitalization
ICU length of stay | 60 days
  ICU length of stay
Brainstem hematoma clearance rate on postoperative days 1, 3, and 7 | 1, 3, and 7 days
  The change in hematoma volume compared to the preoperative CT scan was assessed 1, 3, and 7 days postoperatively.
Incidence of related complications within 14 days, including pneumonia, aphasia, seizures, and lower-extremity deep vein thrombosis | 14 days
  Incidence of related complications within 14 days, including pneumonia, aphasia, seizures, and lower-extremity deep vein thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Yanbing Yu, M.D., Study Chair — China-Japan Friendship Hospital
Locations (3):
- China (3):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Aerospace Center Hospital, Beijing, Beijing Municipality
  - Hebei Provincial People's Hospital, Shijiazhuang, Hebei

IPD SHARING:
Plan to Share IPD: No
The study has not yet begun; we will decide once recruitment starts.

REFERENCES:
- [Background] Lui TN, Fairholm DJ, Shu TF, Chang CN, Lee ST, Chen HR. Surgical treatment of spontaneous cerebellar hemorrhage. Surg Neurol. 1985 Jun;23(6):555-8. doi: 10.1016/0090-3019(85)90002-3. PMID 3992454